CLINICAL TRIAL: NCT03917758
Title: Assessment of the Renin-angiotensin-aldosterone System (RAAS) and Antidiuretic Function in Patients With Type 2 Diabetes Before and During Treatment With Sodium-glucose Co-transporter 2 Inhibitors (SGLT2i): the GliRACo 1 Study
Brief Title: Antidiuretic Function Before and During Treatment With SGLT2 Inhibitors
Acronym: GliRACo1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mauro Maccario, Medical Doctor, Professor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GliRACo 1
Record Dates: First submitted 2019-04-07; First posted 2019-04-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Arterial Hypertension; Body Weight Changes
Keywords: Sodium-Glucose Transporter 2 Inhibitors; Renin-Angiotensin System; Vasopressin; Natriuretic Peptide, Brain; Blood Pressure; Body Composition; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Body Weight Changes; Diabetes Insipidus | interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diabetic patients (Experimental): 30 diabetic patients candidate to treatment with SGLT2i in add-on to metformin.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Start of the treatment with SGLT2i.
  Other Names: Dapagliflozin, Empagliflozin, Canagliflozin

SUMMARY:
Subjects treated with Canagliflozin, Dapagliflozin and Empagliflozin obtained improvement on blood pressure values, body weight and cardiovascular mortality but pathophysiological explanations of these effects are not yet known.

DETAILED DESCRIPTION:
The pathophysiological explanations of the cardiovascular improvement of patients treated with SGLT2i are not yet known: osmotic diuresis and natriuresis, direct effects of weight reduction, increased in nitric oxide release, oxidative stress reduction, local renin-angiotensin-aldosterone system (RAAS) inhibition are the supposed mechanism. In the Literature the diuretic effect of SGLT2i therapy seems to be even stronger than thiazide or thiazide-like drugs. However, it is not defined the role of SGLT2i on antidiuretic function (RAAS, brain natriuretic peptide-BNP and antidiuretic hormone-ADH). Defining this relation could be important for:

* knowing effect of SGLT2i on RAAS (drugs interferences are important particularly during case detection of primary aldosteronism);
* discovering antidiuretic response to SGLT2i treatment and interactions between RAAS, BNP and ADH on the volume improvement induced by this new antidiabetic drugs.

In addition the aim of the study is to define effect of treatment on blood pressure and body composition.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients;
* clinical indication to SGLT2i therapy.

Exclusion Criteria:

* signs and symptoms of poor glycemic control (polydipsia, polyuria and weight loss);
* HbA1c >10% or 86 mmol/mol;
* Body Mass Index (BMI) > 40 Kg/m2;
* personal history of primary and secondary aldosteronism;
* personal history of heart failure;
* personal history of acute kidney injury;
* personal history of chronic kidney disease;
* personal history of liver cirrhosis;
* personal history of protein-wasting syndrome;
* personal history of renin secreting tumor;
* personal history of diabetes insipidus;
* personal history of syndrome of inappropriate antidiuresis (SIAD);
* personal history of hypocortisolism and hypercortisolism;
* therapy with Angiotensin Converting Enzyme inhibitors;
* therapy with Angiotensin Receptor Blockers;
* therapy with renin inhibitors;
* therapy with beta-blockers;
* therapy with alfa2-receptors agonists;
* therapy with Calcium Channel Blockers;
* therapy with diuretics;
* therapy with mineralocorticoid receptor antagonists;
* therapy with non steroidal and steroidal anti-inflammatory drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of antidiuretic function parameters (BNP) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Blood samples for BNP (pg/mL).
Changes from baseline of antidiuretic function parameters (BNP) | 90 days after starting SGLT2i therapy
  Blood samples for BNP (pg/mL).
Changes from baseline of antidiuretic function parameters (vasopressin) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Blood samples for Copeptin (pmol/L).
Changes from baseline of antidiuretic function parameters (vasopressin) | 90 days after starting SGLT2i therapy
  Blood samples for Copeptin (pmol/L).
Changes from baseline of antidiuretic function parameters (osmolality) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Samples for plasma osmolality (mOsm/Kg).
Changes from baseline of antidiuretic function parameters (osmolality) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Samples for urinary osmolality (mOsm/Kg).
Changes from baseline of antidiuretic function parameters (osmolality) | 90 days after starting SGLT2i therapy
  Samples for plasma osmolality (mOsm/Kg).
Changes from baseline of antidiuretic function parameters (osmolality) | 90 days after starting SGLT2i therapy
  Samples for urinary osmolality (mOsm/Kg).
Changes from baseline of antidiuretic function parameters (sodium balance) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Samples for serum sodium (mmol/L).
Changes from baseline of antidiuretic function parameters (sodium balance) | 90 days after starting SGLT2i therapy
  Samples for serum sodium (mmol/L).
Changes from baseline of antidiuretic function parameters (sodium balance) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Samples for urinary sodium (mmol/L).
Changes from baseline of antidiuretic function parameters (sodium balance) | 90 days after starting SGLT2i therapy
  Samples for urinary sodium (mmol/L).
Changes from baseline of antidiuretic function parameters (potassium balance) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Samples for serum potassium (mmol/L).
Changes from baseline of antidiuretic function parameters (potassium balance) | 90 days after starting SGLT2i therapy
  Samples for serum potassium (mmol/L).
Changes from baseline of antidiuretic function parameters (potassium balance) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Samples for urinary potassium (mmol/L).
Changes from baseline of antidiuretic function parameters (potassium balance) | 90 days after starting SGLT2i therapy
  Samples for urinary potassium (mmol/L).
Changes from baseline of renin-angiotensin-aldosterone system parameters (renin) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Blood samples for plasma renin activity (ng/mL/h).
Changes from baseline of renin-angiotensin-aldosterone system parameters (renin) | 90 days after starting SGLT2i therapy
  Blood samples for plasma renin activity (ng/mL/h).
Long term changes from baseline of renin-angiotensin-aldosterone system parameters aldosterone) | Before starting SGLT2i and 30 days the starting SGLT2i therapy
  Blood samples for aldosterone (pg/mL).
Long term changes from baseline of renin-angiotensin-aldosterone system parameters | 90 days after starting SGLT2i therapy
  Blood samples for plasma renin activity (ng/mL/h) and aldosterone (pg/mL)

SECONDARY OUTCOMES:
Changes from baseline of blood pressure values (ABPM) | Before starting SGLT2i and 90 days after the starting
  Mean Systolic and Diastolic Blood Pressure (mmHg)
Changes from baseline of body composition | Before starting SGLT2i and 90 days after the starting
  Variation of parameters of Bioelectrical Impedance Analysis (BIA)
Changes in basal glicemic control | Before starting SGLT2i and 90 days after the starting
  Blood samples for basal glucose (mg/dL).
Changes in long term glicemic control | Before starting SGLT2i and 90 days after the starting
  Blood samples for Glycated albumin (mmol/mol).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro M Maccario, MD, Principal Investigator — Endocrinology, Diabetology and Metabolism; University of Turin; Ezio E Ghigo, MD, Study Chair — Endocrinology, Diabetology and Metabolism; University of Turin
Locations (1):
- Mauro Maccario, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reed JW. Impact of sodium-glucose cotransporter 2 inhibitors on blood pressure. Vasc Health Risk Manag. 2016 Oct 27;12:393-405. doi: 10.2147/VHRM.S111991. eCollection 2016. PMID 27822054
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Lambers Heerspink HJ, de Zeeuw D, Wie L, Leslie B, List J. Dapagliflozin a glucose-regulating drug with diuretic properties in subjects with type 2 diabetes. Diabetes Obes Metab. 2013 Sep;15(9):853-62. doi: 10.1111/dom.12127. Epub 2013 Jun 5. PMID 23668478
- [Result] Shin SJ, Chung S, Kim SJ, Lee EM, Yoo YH, Kim JW, Ahn YB, Kim ES, Moon SD, Kim MJ, Ko SH. Effect of Sodium-Glucose Co-Transporter 2 Inhibitor, Dapagliflozin, on Renal Renin-Angiotensin System in an Animal Model of Type 2 Diabetes. PLoS One. 2016 Nov 1;11(11):e0165703. doi: 10.1371/journal.pone.0165703. eCollection 2016. PMID 27802313
- [Result] Cherney DZ, Perkins BA, Soleymanlou N, Maione M, Lai V, Lee A, Fagan NM, Woerle HJ, Johansen OE, Broedl UC, von Eynatten M. Renal hemodynamic effect of sodium-glucose cotransporter 2 inhibition in patients with type 1 diabetes mellitus. Circulation. 2014 Feb 4;129(5):587-97. doi: 10.1161/CIRCULATIONAHA.113.005081. Epub 2013 Dec 13. PMID 24334175
- [Result] Boertien WE, Riphagen IJ, Drion I, Alkhalaf A, Bakker SJ, Groenier KH, Struck J, de Jong PE, Bilo HJ, Kleefstra N, Gansevoort RT. Copeptin, a surrogate marker for arginine vasopressin, is associated with declining glomerular filtration in patients with diabetes mellitus (ZODIAC-33). Diabetologia. 2013 Aug;56(8):1680-8. doi: 10.1007/s00125-013-2922-0. Epub 2013 Apr 28. PMID 23624546
- [Result] Nogueira-Silva L, Blanchard A, Curis E, Lorthioir A, Zhygalina V, Bergerot D, Baron S, Amar L, Bobrie G, Plouin PF, Menard J, Azizi M. Deciphering the Role of Vasopressin in Primary Aldosteronism. J Clin Endocrinol Metab. 2015 Sep;100(9):3297-303. doi: 10.1210/JC.2015-2007. Epub 2015 Jul 10. PMID 26161452
- [Result] Pikkemaat M, Melander O, Bengtsson Bostrom K. Association between copeptin and declining glomerular filtration rate in people with newly diagnosed diabetes. The Skaraborg Diabetes Register. J Diabetes Complications. 2015 Nov-Dec;29(8):1062-5. doi: 10.1016/j.jdiacomp.2015.07.006. Epub 2015 Jul 9. PMID 26321369
- [Result] DeFronzo RA, Hompesch M, Kasichayanula S, Liu X, Hong Y, Pfister M, Morrow LA, Leslie BR, Boulton DW, Ching A, LaCreta FP, Griffen SC. Characterization of renal glucose reabsorption in response to dapagliflozin in healthy subjects and subjects with type 2 diabetes. Diabetes Care. 2013 Oct;36(10):3169-76. doi: 10.2337/dc13-0387. Epub 2013 Jun 4. PMID 23735727
- [Derived] Berton AM, Parasiliti-Caprino M, Prencipe N, Bioletto F, Lopez C, Bona C, Caputo M, Rumbolo F, Ponzetto F, Settanni F, Gasco V, Mengozzi G, Ghigo E, Grottoli S, Maccario M, Benso AS. Copeptin adaptive response to SGLT2 inhibitors in patients with type 2 diabetes mellitus: The GliRACo study. Front Neurosci. 2023 Mar 20;17:1098404. doi: 10.3389/fnins.2023.1098404. eCollection 2023. PMID 37021137